CLINICAL TRIAL: NCT04438135
Title: Children With Aluminium Contact Allergy: Cutaneous Exposure Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Allergy Research Center, Denmark (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: H-20009217
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2020-06

CONDITIONS: Contact Dermatitis; Contact Allergy; Aluminum Allergy
Keywords: vaccination granuloma; aluminium contact allergy; children; contact dermatitis; repeated open application test; patch test
MeSH Terms: conditions — Dermatitis, Contact; Dermatitis, Allergic Contact

STUDY DESIGN:
Intervention Model Description: Repeated Open Application test
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active test (Active Comparator)
  Interventions: Other: Repeated open application test
- placebo test (Placebo Comparator)
  Interventions: Other: Repeated open application test

INTERVENTIONS:
Other: Repeated open application test — parallel application of two different types of lotion with and without aluminium.

SUMMARY:
Aluminium is used in many different cosmetic products, including make-up, deodorants and sunscreen. The purpose of this study is to investigate whether these everyday skin products with small amounts of aluminium can cause skin reactions in children diagnosed with contact allergy to aluminium.

The study is conducted as a Repeated Open Application Test study (ROAT), a method originally developed to clarify the clinical relevance of questionable and positive patch samples, by imitating everyday use of a skin product.

DETAILED DESCRIPTION:
The study is conducted as a Repeated Open Application Test study (ROAT), a method originally developed to clarify the clinical relevance of questionable and positive patch samples, by imitating everyday use of a skin product.

The skin products will consist of ordinary sunscreens with and without aluminium, with colour code red and blue, respectively (masked for both investigator and participants). At the beginning of the trial, the study participants will be given the two creams. On the lower back of the children, two areas each 10 cm2 are marked with red and blue, respectively. In each area, sunscreen corresponding to the generally recommended amounts must be applied twice a day.

The children should be seen on day 0 for interviews and objective examination. They must then be seen again on day 7 and day 14. On day 14 of the ROAT, a patch test is made to validate the results of the ROAT study. The study is scheduled to last for a maximum of 21 days with 4-5 consultations per child. If there is a skin reaction in connection with the ROAT study before the 14 days have elapsed, the study will end and a patch test will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Children with contact allergies to aluminium, demonstrated by patch tests at the Skin and Allergy Department, Gentofte Hospital and thus registered in the Clinical Database for Contact Allergy.
* Activity (itching) of the granulom within the last six months
* Written consent obtained from all custodians.
* Self-assessed worsening of skin symptoms after contact with aluminium-containing sunscreens.

Exclusion Criteria:

* Treatment with systemic steroid preparations within 1 week.
* Treatment with topical steroid preparations at or near the test area within 1 week.
* Treatment with systemic immune suppression.
* Treatment with antibiotics within 1 week.
* If the children become ill during the study, they should contact the project manager who will clinically assess the child and evaluate whether the child can continue to participate in the study or should be excluded due to the possibility of misinterpretation of any rash.
* Active eczema or other skin symptoms on the tested area

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2022-04-07 (Actual); Study Completion 2022-04-07 (Actual)

PRIMARY OUTCOMES:
positive test | two weeks
  After two weeks of daily application, both test sites on all children will be evaluated and scored according to ROAT guidelines. The ROAT will be considered positive at a score of 5 points or more. Photographs will be taken of all reactions (positive and negative) for documentation.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne Duus Johansen, Prof., Study Director — National Allergy Research Centre
Locations (1):
- National Allergy Research Centre, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No